CLINICAL TRIAL: NCT02835924
Title: A Randomized Phase 2 Study Comparing Different Dose Approaches of Induction Treatment (First Cycle) of Regorafenib in Metastatic Colorectal Cancer (mCRC) Patients
Brief Title: Study Comparing Different Dose Approaches of Induction Treatment of Regorafenib in MCRC
Acronym: RE-ARRANGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-16-01
Record Dates: First submitted 2016-07-08; First posted 2016-07-18 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: regorafenib; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Active Comparator): 160 mg/day 3w on/1w off
  Interventions: Drug: Regorafenib
- Arm B (Experimental): 120 mg/day 3w on/1w off 1st cycle; 160 mg/day 3w on/1w off 2nd cycle on
  Interventions: Drug: Regorafenib
- Arm C (Experimental): 160 mg/day 1w on/1w off 1st cycle; 160 mg/day 3w on/1w off 2nd cycle on
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib

SUMMARY:
The purpose of this study is to assess the safety and tolerability of different dose-escalation approaches of regorafenib in mCRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (IC) obtained before any study specific procedures. Subjects must be able to understand and willing to sign a written informed consent.
2. Male or female subjects 18 years of age.
3. Life expectancy of at least 3 months.
4. Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
5. Measurable metastatic stage IV disease with at least 1 measurable metastatic lesion following RECIST criteria v 1.1.
6. Subjects with metastatic colorectal cancer (Stage IV).
7. Progression during or within 3 months following the last administration of approved standard therapies which must include fluoropyrimidine, oxaliplatin, irinotecan, an anti-VEGF and an anti-EGFR (if RAS WT)
8. Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy
9. Subjects who progress more than 6 months after completion of oxaliplatin containing adjuvant treatment must be retreated with oxaliplatin-based therapy to be eligible. Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study
10. ECOG Performance Status of 0 or 1(within 14 days prior to the initiation of study treatment)
11. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

    * Total bilirubin =1.5 x the upper limit of normal (ULN).
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) = 2.5 x ULN (5 x ULN for subjects with liver involvement of their cancer).
    * Alkaline phosphatase limit = 2.5 x ULN (5 x ULN for subjects with liver and/or bone involvement of their cancer).
    * Lipase = 1.5 x the ULN.
    * Serum creatinine 1.5 x the ULN or = 30 mL/min as calculated using the Cockcroft-Gault equation.
    * Platelet count >100000/mm3, hemoglobin >9 g/dL, absolute neutrophil count (ANC) >1500/mm3.
    * International normalized ratio (INR)/ Partial thromboplastin time (PTT) 1.5 x ULN. (Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard.
    * Blood transfusion to meet the inclusion criteria will not be allowed.
12. Women of childbearing potential and men must agree to use adequate contraception before entering the program until at least 8 weeks after the last study drug administration. The investigator or a designated associate is requested to advise the subject on how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care. Women of childbearing potential must have a blood or urine pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment.

Exclusion Criteria:

1. Prior treatment with regorafenib.
2. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study drug
3. Pregnant or breast-feeding subjects:
4. Congestive heart failure = New York Heart Association (NYHA) class 2.
5. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months).
6. Myocardial infarction less than 6 months before start of study drug.
7. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
8. Uncontrolled hypertension. (Systolic blood pressure > 140 mmHg or diastolic pressure >90 mmHg despite optimal medical management).
9. Arterial or venous thromboembolism within 6 months prior to randomization.
10. Pleural effusion or ascites that causes respiratory compromise (CTCAE Grade 2 dyspnea).
11. Ongoing infection > Grade 2 CTCAE v. 4.0.
12. Known history of human immunodeficiency virus (HIV) infection.
13. Known history of active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
14. Subjects with seizure disorder requiring medication.
15. History of organ allograft.
16. Subjects with evidence or history of any bleeding diathesis, irrespective of severity.
17. Any hemorrhage or bleeding event = CTCAE Grade 3 within 4 weeks prior to the start of study medication.
18. Non-healing wound, ulcer, or bone fracture.
19. Renal failure requiring hemo-or peritoneal dialysis.
20. Dehydration CTCAE v. 4.0 Grade = 1.
21. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
22. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
23. Any illness or medical conditions that are unstable or could jeopardize the safety of the subject and his/her compliance in the study.
24. Interstitial lung disease with ongoing signs and symptoms
25. Persistent proteinuria of CTCAE Grade 3 (>3.5g/24 hours).
26. Subjects unable to swallow oral medications.
27. Any malabsorption condition.
28. Unresolved toxicity higher than CTCAE (v. 4.0) > Grade 1 attributed to any prior therapy/procedure excluding alopecia, hypothyroidism and oxaliplatin induced neurotoxicity > Grade 2.
29. Subjects treated with strong CYP3A4 inhibitors or inducers (refer to appendix 8 and to section 6.3.8. Prohibited concomitant medication).
30. Subjects receiving G-CSF within 3 weeks prior to signing the ICF
31. Concomitant participation or participation within the last 30 days in another clinical trial
32. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 weeks (or within 6 weeks for mitomycin C) before starting to receive study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with G3/G4 treatment-related AEs in each arm according to CTCAE v4.03 criteria. | 30 months

SECONDARY OUTCOMES:
Percentage of total administrated dose over the planned dose accomplished in each arm. | 30 months
Dose intensity during the whole treatment. | 30 months
Dose intensity during first two cycles. | 2 months
Disease control rate (DCR) | 30 months
Progression-free survival (PFS) | 30 months
Time to treatment failure (TTF) | 30 months
Overall survival (OS) | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Argiles, Study Chair — Hospital Universitary Vall d'Hebron; Josep Mª Tabernero, MD-PhD, Study Chair — Hospital Universitary Vall d'Hebron
Locations (1):
- Spanish Cooperative Group for the Treatment of Digestive Tumors, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Argiles G, Mulet N, Valladares-Ayerbes M, Vieitez JM, Gravalos C, Garcia-Alfonso P, Santos C, Tobena M, Garcia-Paredes B, Benavides M, Cano MT, Loupakis F, Rodriguez-Garrote M, Rivera F, Goldberg RM, Cremolini C, Bennouna J, Ciardiello F, Tabernero JM, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD) and UNICANCER GI; The, REARRANGE investigators; Principal investigator; Argiles G, Tabernero J; Steering Committee; Investigators. A randomised phase 2 study comparing different dose approaches of induction treatment of regorafenib in previously treated metastatic colorectal cancer patients (REARRANGE trial). Eur J Cancer. 2022 Dec;177:154-163. doi: 10.1016/j.ejca.2022.09.037. Epub 2022 Oct 14. PMID 36335783
- [Derived] Weinberg BA, Hartley ML, Salem ME. Precision Medicine in Metastatic Colorectal Cancer: Relevant Carcinogenic Pathways and Targets-PART 2: Approaches Beyond First-Line Therapy, and Novel Biologic Agents Under Investigation. Oncology (Williston Park). 2017 Jul 15;31(7):573-80. PMID 28712102